CLINICAL TRIAL: NCT04487197
Title: SARS-CoV2 (COVID-19) Seroepidemiological Investigation in Transplanted Population Subjects of Kidney, Kidney-pancreas, Isolated Pancreas, Langerhans Islets
Brief Title: SARS-CoV2 (COVID-19) Seroepidemiological Transplanted Subjects (Kidney, Kidney-pancreas, Pancreas, Langerhans Islets)
Status: Completed | Type: Observational
Sponsor: Antonio Secchi (Other)
Responsible Party: Sponsor-Investigator, Antonio Secchi, MD, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: COVID-SIERO TRAPIANTI
Record Dates: First submitted 2020-07-24; First posted 2020-07-27 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Kidney Transplant; Pancreatic Transplat; Pancreatic Islets Langerhans
Keywords: COVID-19 infection; Transplanted patients; kidney transplants; pancreas transplants; pancreatic islet transplantation
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: * Adult patients (age ≥ 18 years),
  * kidney or pancreas or pancreatic islets transplantation
  * transplanted patients (period: 01.01.2020 to 30.06.2020)
  Interventions: Procedure: blood sample for seroepidemiological investigation
- Cohort 2: * Adult patients (age ≥ 18 years),
  * kidney or pancreas or pancreatic islets transplantation
  * Transplanted patients in follow-up since 01.01.2020 or trasplanted patients after 30.06.2020.
  Interventions: Procedure: blood sample for seroepidemiological investigation

INTERVENTIONS:
Procedure: blood sample for seroepidemiological investigation — blood sample for seroepidemiological investigation

SUMMARY:
Evaluate SARS-CoV2 infection and the degree of immunity possibly developed in transplanted population using the Luciferase Immuno Precipitation System (LIPS) test.

ELIGIBILITY:
Inclusion Criteria Cohort 1:

* Adult patients (age ≥ 18 years),
* Kidney or pancreas or pancreatic islets transplantation
* Transplanted patients (period: 01.01.2020 to 30.06.2020)
* Informed Consent signed

Inclusion Criteria Cohort 2:

* Adult patients (age ≥ 18 years),
* Kidney or pancreas or pancreatic islets transplantation
* transplanted patients in follow-up since 01.01.2020 or trasplanted patients after 30.06.2020.
* Informed Consent signed

Exclusion Criteria both Cohort (1&2):

Symptomatology such as fever> 37.5, and / or cough and / or respiratory distress and / or diarrhea / vomiting in 14 days prior to collection of blood sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transplanted Kidney, Pancreas or Pancreatic Islet patients
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Serum-prevalence of COVID-19 TX | From 15 July 2020 to 15 January 2021
  Evaluation of serum-prevalence data transplanted patients (symptomatic vs asymptomatic patients)
Serum-prevalence of COVID-19 / Age, Gender, Type of transplantation, comorbities, Italian regions-proviences transplanted patients | From 15 July 2020 to 15 January 2021
  Correlation serum-prevalence of COVID-19 / Age, Gender, Type of transplantation, comorbities, Italian regions-proviences transplanted patients

SECONDARY OUTCOMES:
Asymptomatic or subclinical infections in transplanted patients | From 15 July 2020 to 15 January 2021
  Determine % Asymptomatic or subclinical infections in transplanted patients
Risk factors for infection COVID-19 transplanted patients | From 15 July 2020 to 15 January 2021
  Determine risk factors for infection COVID-19 (comparison symtomatic and asymtomatic transplanted patients)
Hospitalization rate COVID-19 transplanted patients | From 15 July 2020 to 15 January 2021
  Evaluate hospitalization rate in transplanted patients
Mortality rate COVID-19 transplanted patients | From 15 July 2020 to 15 January 2021
  Evaluate mortality rate in transplanted patients

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided